CLINICAL TRIAL: NCT07102667
Title: The Optimal Protein Intake to Enhance Muscle Mass in Elderly Patients With Pre-dialysis Chronic Kidney Disease: A Randomized Active-Controlled Trial
Brief Title: The Optimal Protein Intake to Enhance Muscle Mass in Elderly Patients With Pre-dialysis Chronic Kidney Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Chawalya Angsuwatjarakorn, MD, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0182/68
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia; Chronic Kidney Disease
Keywords: Sarcopenia; Chronic kidney disease; Protein intake; Nutrition
MeSH Terms: conditions — Sarcopenia; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein intake of 1.2 g/kg/day (Experimental)
  Interventions: Behavioral: Protein intake 1.2 g/kg/day and resistance exercise
- Protein intake of 1.0 g/kg/day (Active Comparator)
  Interventions: Behavioral: Protein intake 1.0 g/kg/day and resistance exercise

INTERVENTIONS:
Behavioral: Protein intake 1.2 g/kg/day and resistance exercise — Protein intake of 1.2 g/kg/day in combination with resistance exercise using resistance bands
  Arms: Protein intake of 1.2 g/kg/day
Behavioral: Protein intake 1.0 g/kg/day and resistance exercise — Protein intake 1.0 g/kg/day in combination with resistance exercise using resistance bands
  Arms: Protein intake of 1.0 g/kg/day

SUMMARY:
The goal of this clinical trial is to determine whether increasing protein intake in elderly adults with pre-dialysis chronic kidney disease, in combination with resistance exercise, improves muscle mass without worsening renal function.The main questions it aims to answer are:

* Does a protein intake of 1.2 g/kg BW/day combined with exercise improve muscle mass better than a protein intake of 1.0 g/kg BW/day?
* Does a protein intake of 1.2 g/kg BW/day combined with exercise lead to greater improvements in muscle strength and function?
* Does a protein intake of 1.2 1.2 g/kg BW/day combined with exercise cause a decline in renal function (eGFR) compared to a protein intake of 1.0 1.2 g/kg BW/day?

Researchers will compare a group assigned to intake 1.2 g/kg BW/day of protein with another group assigned to intake 1.0 g/kg BW/day, to assess whether the higher intake improves muscle mass and physical performance without causing harm.

Participants will

* be assessed for body composition, physical performance and nutritional intake.
* be assigned to consume protein at either 1.2 or 1.0 g/kg/day.
* perform a home-based resistance exercise program using resistance bands.
* provide blood and urine sample to monitor renal function.
* visit the clinic at weeks 12 and 24 for repeated measurement.

ELIGIBILITY:
Inclusion Criteria:

* Thai adults aged ≥ 65 years
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) 30-59 ml/min/1.73 m2
* Sarcopenia or presarcopenia (diagnosis based on Asian Working Group for Sarcopenia (AWGS) 2019 definition)

Exclusion Criteria:

* Active cardiopulmonary disease(s) or uncontrolled hypertension with contraindications to resistance training
* Physically or cognitively unable to participate in the resistance exercise program (e.g. dementia), as determined by the attending physician
* Limitations of body measurements and interpretation using Bioelectrical Impedance Analysis (BIA) e.g. presence of pacemaker, surgical metal implants
* Meets the definition of AKI or AKD, defined as alterations in kidney function within the past 3 months
* Severe vitamin D deficiency (25-OH Vitamin D level < 10 ng/mL)
* Refuses to give consent to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Between-Group Differences in Muscle Mass Changes at 6 Months | From enrollment to the end of intervention at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand